CLINICAL TRIAL: NCT07147699
Title: Evaluation of the Effectiveness of the CardioStory Device in Distinguishing Heart Failure From Other Causes in Patients Presenting With Dyspnea
Acronym: CARDIOSTORY
Status: Not yet recruiting | Type: Observational
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, professor, Hôpital Universitaire Sahloul
Other Study IDs: CARDIOSTORY
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Dyspnea; Heart Failure Acute
Keywords: dyspnea; acute heart failure
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: cardiostory — measure the pressure of remplissage

SUMMARY:
The CARDIOSTORY.TN study is a prospective observational study at Sahloul University Hospital (Sousse, Tunisia) evaluating the CardioStory device for distinguishing heart failure (HF) from other causes of acute dyspnea.

Background: Dyspnea is common in emergencies, and differentiating cardiac from non-cardiac causes is often delayed by the limits of echocardiography and BNP tests. CardioStory is a rapid (~2 minutes), non-invasive tool that measures cardiac filling pressure, a key HF marker.

Objectives:

Primary: Assess CardioStory's diagnostic accuracy.

Secondary: Compare it with echocardiography and NT-proBNP, evaluate ease of use, and measure time to diagnosis.

Methods:

Adults (≥18) with acute dyspnea (<7 days) included; unstable or traumatic/allergic cases excluded.

CardioStory results will be compared to standard diagnostics.

Sample size: 850 patients over 12 months.

Outcome: If accurate, CardioStory could be a fast, practical diagnostic tool for emergency settings.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years

  * Recent onset dyspnea (less than 7 days)
  * Informed consent obtained

Exclusion Criteria:

* • Age inferior to 18 years,

  * Severe comorbidity, hemodynamic compromise or immediate need for mechanical ventilation were exclusion criteria.
  * Dyspnea clearly of traumatic or allergic origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: every patient consulting with dyspnea
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the CardioStory device in identifying heart failure (sensitivity, specificity, PPV, NPV). | 12 hours

SECONDARY OUTCOMES:
o Concordance between CardioStory and standard diagnostic tools o Time to diagnosis o Ease of use and practicality (via physician questionnaire) | 12 hours